CLINICAL TRIAL: NCT02853656
Title: Time to Delivery of Preterm Birth
Status: Terminated | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B868; 194502 (Other: IRAS ID)
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Pre Term Birth
Keywords: preterm birth; gestation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Preterm birth (babies being born before 34 weeks pregnancy) occurs in approximately 11% of pregnancies; preterm birth can lead to complications for the baby.

When mothers are identified as being at risk of going into preterm birth (giving birth within the next 14 days) there are several treatments available that may help reduce the likelihood of complications for the baby. These treatments usually need to be started within 24 hours so it is very important that diagnosing preterm labour in not only fast but accurate.

There are several methods commonly used within hospitals for diagnosing mothers who may be at risk of going into preterm labour. The two most common ones are foetal fibronectin (fFN) and phosphorylated insulin-like growth factor binding protein 1 (phIGFBP-1).

The purpose of this study is to compare the two tests to see which is more accurate at predicting preterm birth.

DETAILED DESCRIPTION:
Preterm birth (babies being born before 34 weeks pregnancy) occurs in approximately 11% of pregnancies; preterm birth can lead to complications for the baby.

When mothers are identified as being at risk of going into preterm birth (giving birth within the next 14 days) there are several treatments available that may help reduce the likelihood of complications for the baby. These treatments usually need to be started within 24 hours so it is very important that diagnosing preterm labour in not only fast but accurate.

There are several methods commonly used within hospitals for diagnosing mothers who may be at risk of going into preterm labour. The two most common ones are foetal fibronectin (fFN) and phosphorylated insulin-like growth factor binding protein 1 (phIGFBP-1).

The purpose of this study is to compare the two tests to see which is more accurate at predicting preterm birth.

This is a prospective comparative study of fFN (control) and PhIGFBP-1 test (comparator) for women with singleton pregnancies between 22-34 weeks gestation presenting with self-reported signs, symptoms or complaints suggestive of preterm labour.

Both tests will be done on every participant - the tests will be sequenced so that every 5 participants the fFN test is undertaken first and then the next cohort of 5 will have the PhIGFBP-1 swab taken first. This is to remove any potential biases surrounding which test was undertaken first. Data collection (case report forms (CRFs)) will clearly document which test was performed 1st and 2nd.

ELIGIBILITY:
Inclusion criteria

* aged ≥ 18 years
* confirmed pregnancy
* gestational age between 22 and 34 weeks
* self-reported signs, symptoms or complaints suggestive of preterm labour;

  * abdominal pain
  * contractions
  * pelvic pressure

Exclusion criteria

* unable to provide written informed consent
* multiple pregnancy
* participating in an interventional clinical trial
* a symptom not associated with idiopathic threatened preterm delivery (e.g. trauma)
* contraindicated to either fFN or PhIGFBP-1; e.g.

  * vaginal bleeding
  * cervical dilation ≥3cm dilated
  * evidence of rupture of membranes
  * had intercourse in last 24 hours
  * cervical cerclage in situ
  * placenta praevia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with singleton pregnancy between 22-34 weeks gestation with signs and symptoms of pre term birth
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
diagnosis of heightened risk of imminent delivery | 7 days
  preterm birth at 7 days
diagnosis of heightened risk of imminent delivery | 14 days
  preterm birth at 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Amaju Ikomi, MBBS FRCOG, Study Director — Basildon and Thurrock University Hospitals NHS FT
Locations (1):
- Basildon Hospital, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No